CLINICAL TRIAL: NCT05451823
Title: A Comparison of Post-auricular and Frontal Bispectral Index Values Obtained During Renal Surgeries
Brief Title: Post-auricular Versus Frontal Bispectral Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amany Faheem, Assistant professor of anesthesiology, intensive care, and pain medicine, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: post-auricular bispectral
Record Dates: First submitted 2022-06-26; First posted 2022-07-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Renal Surgeries
Keywords: frontal bispectral index; post-auricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post auriclar-frontal (Experimental): Frontal sensors will be applied with lead 1 at the center of the forehead; lead 2, 2.8 cm lateral to lead 1; and lead 3 at the temporal area between the lateral canthus and the hairline.
  Post auriclar sensors will be applied to the same side of the face, with lead 1 approximately 2.5 cm medial to the mastoid area, post-auricularly next to the hairline. Lead 2 will be attached at the mastoid area and lead 3 will be attached on the same side at the temporal area between the lateral canthus and the hairline.
  Interventions: Device: Post auriclar-frontal

INTERVENTIONS:
Device: Post auriclar-frontal — Frontal sensors will be applied with lead 1 at the center of the forehead; lead 2, 2.8 cm lateral to lead 1; and lead 3 at the temporal area between the lateral canthus and the hairline.
  Post auriclar sensors will be applied to the same side of the face, with lead 1 approximately 2.5 cm medial to the mastoid area, post-auricularly next to the hairline. Lead 2 will be attached at the mastoid area and lead 3 will be attached on the same side at the temporal area between the lateral canthus and the hairline.

SUMMARY:
Electroencephalogram (EEG) derived monitors during practice of general anesthesia; allow the titration and maintenance of an adequate depth of anesthesia, advantages from reducing the recovery time after waking, as well as the risk of anesthetics adverse events .

There are various types of EEG-derived monitoring devices that are used to monitor the depth of anesthesia, and among the established devices is bispectral index (BIS) monitor. It is a quantitative electroencephalographic device that is widely used to assess the hypnotic component of anesthesia, and a level between 40 and 60 is recommended for an adequate level of the hypnotic state.

However, the use of BIS in certain surgeries is challenging because of the proximity of the forehead sensor to the surgical site. There are high possibilities of interruption of BIS recording due to contamination of the forehead sensor with blood or antiseptic cleaning solution. At the same time, the design and size of a BIS forehead sensor in the form of a long strip can also interfere with the site of surgical incision.

Several alternative BIS sensor placements have been studied for cases in which the frontal setup is not feasible. However, few studies studied the placement of the BIS sensor at the post-auricular area as an alternative method of monitoring the depth of anesthesia.

DETAILED DESCRIPTION:
Twelve Patients age ≥18 years, ASA I-III patients scheduled for elective renal surgeries.

Monitoring of the depth of anesthesia will be performed using an Inﬁnity BISx SmartPod® (Aspect Medical Systems, Newton, MA, USA) and an Inﬁnity® Delta XL monitor (Dräger Medical, Lübeck, Germany). Two standard BISx Quatro® Sensors (Aspect Medical Systems) were placed at the forehead and post-auricular area.

Before the induction of anesthesia, 2 BIS sensors (BISTM Quatro Sensors, Aspect Medical Systems, Newton, MA, USA) will be applied to each patient, 1 across the forehead and 1 along the post auricular area and attached each sensor to each BIS monitor (BIS-VistaTM monitors, Aspect Medical Systems, Newton, MA, USA).

During induction, patients will be instructed to keep their faces relaxed (eyes closed, mouth closed, no facial expressions).

The skin on the forehead will be cleaned with an alcohol 70% swab, and 2 to 5 seconds of digital pressure applied over the sensor leads. The sensor is comprised of disposable wet gel electrodes. Electromyographic activity of the frontalis muscle is measured by lead 4, which is the ground electrode as well.

Frontal sensors will be applied with lead 1 at the center of the forehead; lead 2, 2.8 cm lateral to lead 1; and lead 3 at the temporal area between the lateral canthus and the hairline.

Post auriclar sensors will be applied to the same side of the face, with lead 1 approximately 2.5 cm medial to the mastoid area, post-auricularly next to the hairline. Lead 2 will be attached at the mastoid area and lead 3 will be attached on the same side at the temporal area between the lateral canthus and the hairline.

The titration of anesthetic depth will be maintained at BIS values between 40-60.

Sudden, high EMG scores were identified as artifacts and the associated BIS values were eliminated in data analysis.

Measurements:

From each BIS monitor, the investigators will collect 3 pieces of data at each of 6 times points: BIS score, signal quality index (SQI) score determining the strength of the signal, and electromyography (EMG) score: before the induction of anesthesia (awake), at loss of the eyelash reflex (LOC), after intubation (intubation), after the first surgical incision (incision), every 30 minutes during the intraoperative period (maintenance), and at spontaneous eye opening upon emergence from anesthesia (emergence).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged≥18 years
* ASA I-III
* patients scheduled for elective renal surgeries

Exclusion Criteria:

* Patients with disabling central nervous system
* cerebrovascular disease
* those currently taking psychiatric medication
* those with a history of neurosurgical intervention
* those with contraindications for the placement of electrodes over forehead and post-auricular area (e.g., having skin infections)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Post-auricular and frontal BIS values | 5 minutes before induction of aneasthesia
  Post-auricular and frontal BIS values

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tantan University Hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelrahman AMF, Elbadry AA, Omara AF. Comparison of post-auricular and frontal bispectral index values obtained during renal surgeries. BMC Anesthesiol. 2023 Dec 19;23(1):417. doi: 10.1186/s12871-023-02372-x. PMID 38114941